CLINICAL TRIAL: NCT05082805
Title: Therapeutic Strategy Concerning the Drug Management Associated With bDMARDs or tsDMARDs in Rheumatoid Arthritis and Psoriatic Arthritis
Brief Title: Therapeutic Strategy Associated With bDMARDs or tsDMARDs in Rheumatoid Arthritis and Psoriatic Arthritis
Acronym: STRATEGE2
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Nordic Pharma SAS (Industry)
Responsible Party: Sponsor
Other Study IDs: STRATEGE 2
Record Dates: First submitted 2019-06-24; First posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a longitudinal, observational, prospective, multicentre study conducted in France, among a representative sample of rheumatology doctors.

The aim of this study is to describe in real life the therapeutic strategy when faced with a patient with rheumatoid arthritis (RA) or psoriatic arthritis (PsA) who requires initiation of treatment with biotherapy or targeted therapy. The evolution of the disease and the possible therapeutic adaptations will then be followed for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Major patient (age ≥ 18 years)
* Patient with RA according to American College of Rheumatology (ACR) / European Congress of Rheumatology (EULAR) 2010 or ACR 1987 or patient with PsA according to ClASsification criteria for Psoriatic ARthritis (CASPAR) criteria
* Patient undergoing treatment with methotrexate (MTX) (oral or injectable) initiated for at least 3 months.
* Naïve patient of biotherapy or tsDMARD and requiring the introduction of a first bDMARD or tsDMARD due to the activity of the disease.
* Patient informed and accepting the computer processing of his/her medical data and informed of his/her rights of access and rectification.

Exclusion Criteria:

* Patient participating in an interventional study in rheumatology
* Patient with axial spondyloarthritis (for patients with PsA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RA or PsA patient undergoing treatment with MTX for at least 3 months and requiring the introduction of a first bDMARD or tsDMARD due to the activity of the disease will be asked to participate from bDMARD or tsDMARD treatment introduction (inclusion visit) up to 24 months after inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-02-25 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The Primary Outcome Measure is not provided for now to the investigators (and public) in order not to bias the therapeutic strategies. | 12 months after inclusion
  Not provided as Outcome 1 is blinded

SECONDARY OUTCOMES:
Main criteria analysis | 24 months after inclusion
  Same Outcome 1, but at 24 month. This outcome is blinded too.
Therapeutic adaptations of conventional synthetic disease-modifying antirheumatic drugs (csDMARDs), biologic DMARDs (bDMARDs), targeted synthetic DMARDs (tsDMARDs), Nonsteroidal anti-inflammatory drugs (NSAIDs) and corticosteroids | 12 and 24 months after inclusion
  delays, changes in dosage, changes in the route of administration, reasons for adaptations ...
Disease outcome | 12 and 24 months after inclusion
  disease activity (Disease Activity Score DAS28 and Disease Activity in PSoriatic Arthritis DAPSA)), percentage of patients in remission, quality of Life (Dermatology Life Quality Index (DLQI))
Patient adherence to treatment | 12 and 24 months after inclusion
  The variation of patients' adherence to antirheumatic treatments evaluated by the Compliance Questionnaire for Rhumatology (CQR19).
Fatigue and pain | 12 and 24 months after inclusion
  Visual Analog Scale (VAS) anchored by 2 verbal descriptors, one for each symptom extreme : 0 (no fatigue, no pain) to 10 (maximum fatigue, maximum pain).
Functional capacity (Health Assessment Questionnaire (HAQ)) | 12 and 24 months after inclusion
  This questionnaire is completed by patients at baseline, 12 months and 24 months.
Cross-perception (doctor / patient) about participation in the "shared medical decision" | 12 and 24 months after inclusion
  This outcome is based on 2 mirror questions (one asked to the physician and on to the patient). They are asked if the decision to adapt the therapeutic decision is a "shared medical decision". Five answers are possible from "fully" to "not at all".
Care path at the end of the visit | 12 and 24 months after inclusion
  The physician is asked about the patient pathway (How and by whom the patient will be followed : nurse, other physicians)

CONTACTS AND LOCATIONS:
Overall Officials: Hélène HERMAN-DEMARS, MD, Study Director — Nordic Pharma; René Marc FLIPO, Prof, Principal Investigator — CHRU LILLE; Cécile GAUJOUX-VIALA, Dr, Principal Investigator — CHU Nîmes; Emmanuelle DERNIS, Dr, Principal Investigator — CH Le Mans; Éric SENBEL, Dr, Principal Investigator — Marseille
Locations (1):
- Nordic Pharma, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaujoux-Viala C, Dernis E, Senbel E, Herman-Demars H, Becker J, Flipo RM. Methotrexate Maintenance After Initiation of Biological or Targeted Synthetic DMARDs in Rheumatoid Arthritis: Results from the 2-Year Longitudinal Prospective Non-interventional STRATEGE2 Study. Rheumatol Ther. 2026 Feb;13(1):157-177. doi: 10.1007/s40744-025-00806-1. Epub 2025 Dec 3. PMID 41335306